CLINICAL TRIAL: NCT04921995
Title: Postponing or Omitting Re-irradiation After Tislelizumab Plus Chemotherapy in Unresectable Recurrent Loco-regionally Advanced Nasopharyngeal Carcinoma
Brief Title: Immunotherapy and Chemotherapy in Unresectable Recurrent Loco-regionally Advanced Nasopharyngeal Carcinoma
Acronym: RETICULA-NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoshen Wang, Director of Department of Radiation Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021052-1
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Nasopharyngeal Carcinoma; Unresectable Nasopharyngeal Carcinoma; Chemotherapy Effect; Immunotherapy; Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Main group: Patients with unresectable, recurrent NPC who were treated with tislelizumab plus investigator's choice chemotherapy, with re-irradiation postponed or omitted. But there are two subgroups, one subgroup was ICI naive patients and were given first line tislelizumab plus investigator's choice chemotherapy. The other subgroup included patients who displayed no response to or progressed after previous PD-1 blockade, and were treated with tislelizumab rechallenge plus either chemotherapy or low dose SBRT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Main group: Patients will be given first line tislelizumab plus investigator's choice chemotherapy, with re-irradiation postponed or omitted.
  Subgroup: For patients that progressed after exposure to another PD-1 antibody, tislelizumab rechallenge combined with either low dose SBRT or low dose gemcitabine and metronomic capecitabine is accepted as a second subgroup.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — 1. Chemotherapy (including but not limited to following):
     GP regimen: gemcitabine 1000mg/m2 d1, d8 + cisplatin 25 mg/m2 d1-3, every 3 weeks for 4-6 cycles; GX regimen: gemcitabine 800mg/m2 d1 + capecitabine 750 mg/m2 d1-14, every 3 weeks for 4-6 cycles.
     Capecitabine: 750 mg/m2 d1-14, every 3 weeks until unacceptable toxicities or patient's withdraw.
  2. anti-PD-1 antibody: Tislelizumab concurrently with chemotherapy: 200mg, every 3 weeks for 12 weeks. Tislelizumab in maintenance period: 200mg every 3 weeks or 400mg every 6 weeks, until one year or disease progression, or in the case of intolerable toxicities.

SUMMARY:
This is an open-label, multi-center, phase II trial to evaluate the safety and efficacy of postponing or omitting re-irradiation after systemic therapy with tislelizumab and chemotherapy in patients with unresectable recurrent loco-regionally advanced nasopharyngeal carcinoma. Patients who did not respond to or progressed on another ICI are allowed to receive tislelizumab rechallenge as a subgroup.

DETAILED DESCRIPTION:
High dose reirradiation is usually recommended for unresectable recurrent loco-regionally advanced nasopharyngeal carcinoma. However, it potentially adds to the RT-related severe toxicities and deaths. This trial aims to investigate the feasibility of postponing or even omitting re-irradiation based on effective first-line systemic therapy with tislelizumab and chemotherapy. For patients that progressed after exposure to another PD-1 antibody,tislelizumab rechallenge is accepted as a second subgroup.In this trial, all patients will receive chemotherapy (on doctors' recommendation) and PD-1 antibody (tislelizumab 200mg every three weeks). Patients with no response to the systemic therapy will receive salvage low dose re-irradiation delivered by SBRT, while those who showed complete or partial response will continue maintenance therapy until progression, death or intolerable toxicity, and reirradiation will be postponed or omitted.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as local recurrence ± regional recurrence after ≥1 year of radical treatment;
2. Not suitable for surgery;
3. Clinical stage rT3-4N0-2 (rII-IVa, AJCC/UICC 8th);or residual disease afer surgery.
4. ECOG score 0-1;
5. No prior treatment to rNPC, such as radiotherapy, chemotherapy, immunotherapy or biotherapy;
6. No contraindications to immunotherapy or chemoradiotherapy;
7. Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;
8. Adequate liver function: ALT/AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;
9. Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
10. Take effective contraceptions during and two months after treatment;
11. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Have local necrosis in recurrent lesions, estimated with bleeding risk;
2. Unexplained fever > 38.5 ℃, except for tumor fever;
3. Treated with ≥ 5 days antibiotics one month before enrollment;
4. Have active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy);
5. Have a known history of human immunodeficiency virus (HIV), active Hepatitis B (HBV-DNA ≥10E3copiers/ml) or hepatitis C virus (HCV) antibody positive;
6. Have ≥G3 late toxicities, except for skin, subcutaneous tissue or mucosa;
7. Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment;
8. Have known allergy to large molecule protein products or any compound of study therapy;
9. Pregnant or breastfeeding;
10. Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
11. Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months
  Defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) .
Progress-free survival (PFS) | 2 year
  Defined from date of enrollment to date of first documentation of progression or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 year
  Defined from date of enrollment to date of first documentation of death from Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Adverse events (AEs) | 2 year
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Quality of life (QoL) | 1 year
  QoL scores were assessed by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshen Wang, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Background] Kong F, Zhou J, Du C, He X, Kong L, Hu C, Ying H. Long-term survival and late complications of intensity-modulated radiotherapy for recurrent nasopharyngeal carcinoma. BMC Cancer. 2018 Nov 20;18(1):1139. doi: 10.1186/s12885-018-5055-5. PMID 30453915
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Liu LT, Chen QY, Tang LQ, Zhang L, Guo SS, Guo L, Mo HY, Zhao C, Guo X, Chen MY, Qian CN, Zeng MS, Hong MH, Shao JY, Sun Y, Ma J, Mai HQ. With or without reirradiation in advanced local recurrent nasopharyngeal carcinoma: a case-control study. BMC Cancer. 2016 Oct 7;16(1):774. doi: 10.1186/s12885-016-2803-2. PMID 27717335